CLINICAL TRIAL: NCT05383469
Title: Comparison of the Efficacy of Active Versus Passive Methods in Patients With Chronic Venous Insufficiency
Brief Title: Efficacy of Active Versus Passive Methods in Chronic Venous Insufficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Saliha Gürdal Karakelle, Research .Assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 99984023-302.14.68-
Record Dates: First submitted 2022-02-09; First posted 2022-05-20 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Chronic Venous Insufficiency
Keywords: exercise; compression; neuromuscular electrical stimulation; massage
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Massage

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Compression Group (Active Comparator): Routine compression therapy will be administered.
  Interventions: Other: Compression Therapy
- Active Group (Experimental): Exercise training will be administered.
  Interventions: Other: Exercise Training; Other: Compression Therapy
- Passive Group (Experimental): Massageand neuromuscular electrical stimulation will be administered.
  Interventions: Other: Massage; Other: Neuromuscular Electrical Stimulation; Other: Compression Therapy

INTERVENTIONS:
Other: Exercise Training — Endurance training with a resistance-free bicycle ergometer Strength training with bodyweight Non-resistance ankle pumping exercises
  Arms: Active Group
Other: Massage — Classical massage including superficial and deep stroking and friction methods for the lower extremity.
  Arms: Passive Group
Other: Neuromuscular Electrical Stimulation — Symmetrical biphasic current at a frequency of 30-85 Hz
  Arms: Passive Group
Other: Compression Therapy — Compression therapy is a treatment applied to patients in the form of Four Layer Compression Bandage and Compression Stocking. Four Layer Compression Bandage is a treatment that requires four different types of bandages. The compression stocking is an elastic stock with various tension and length.

SUMMARY:
The aim of our study was to compare the effectiveness of active and passive practices in patients with CVI.

DETAILED DESCRIPTION:
Volunteers who have been diagnosed with venous insufficiency according to the criteria of inclusion, who applied to Cardiovascular Surgery Department will be included this study.

Participants will be randomly allocated 3 groups using the 'Research Randomizer' website. In all groups, a common evaluation protocol will be applied to the patients.

Compression therapy will be applied to the first group. Active treatment in addition to compression therapy will be applied to the second group. Passive treatment in addition to compression therapy will be applied to the third group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of venous insufficiency with duplex ultrasonography
* Classification of CEAP (Clinical-Etiological-Anatomical-Pathological) used in venous insufficiency is C3-C4-C5-C6
* Ankle-brachial index (ABI) is less than 0.7
* Possibility to communicate in written and verbal in Turkish
* Have a level of cognitive ability to understand the instructions given

Exclusion Criteria:

* Presence of deep vein thrombosis
* Ulceration or open burn wound in lower extremity greater than 4 cm
* Presence of infected ulceration
* Cardiorespiratory insufficiency
* Orthopedic, rheumatologic or neurological comorbidities restrain the exercise in the lower extremity
* Presence of a psychiatric illness requiring the use of prescribed medicines

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2022-12-25 (Actual); Study Completion 2023-09-02 (Actual)

PRIMARY OUTCOMES:
Circumference measurements | Change from Baseline circumferences at 8 weeks.
  Circumference measurements will be recorded at 4 cm intervals to evaluated to edema.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | Assessment will be performed at baseline and at 8 weeks.
  The levels of pain felt rest/activity/night will be measured using visual analogue scale (VAS). Patients will be asked to evaluate their pain status with a 10-point scale and high scores are positively correlated with pain.
Venous Clinical Severity Score (VCSS) | Assessment will be performed tat baseline and at 8 weeks.
  Clinical severity will be measured by Venous Clinical Severity Score (VCSS).The VCSS was subsequently developed as an evaluative instrument that would be responsive to changes in disease severity over time and in response to treatment.The total score is at least 0 and at most 30, and the low scores are positively correlated with the severe clinical condition.
Handheld Dynamometer | Assessment will be performed at baseline and at 8 weeks.
  The muscle strength of the gastrocnemius and tibialis anterior muscles will be evaluated using the handheld dynamometer.
6-Minute Walking Test | Assessment will be performed at baseline and at 8 weeks.
  Functional capacity will be evaluated with the 6-minute walking test. The 6-minute walking test (6 MWT) is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes.
10-Meter Walking Test | Assessment will be performed at baseline and at 8 weeks.
  Walking speed will be evaluated with the 10-meter walking test. 10-meter walking test is used to assess walking speed in meters/second (m/s) over a short distance.
Chronic Venous Disease Quality of Life Questionnaire (CIVIQ) 20 | Assessment will be performed at baseline and at 8 weeks.
  Quality of Life will be evaluated with the Chronic Venous Disease Quality of Life Questionnaire (CIVIQ) 20. CIVIQ 20 is a disease-related quality of life assessment form especially for chronic venous insufficiency patients. The total score is at least 0 and at most 100, and the higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Büyükçekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No